CLINICAL TRIAL: NCT00504231
Title: Intradermal vs. Intramuscular Delivery of Influenza Vaccine in Immunocompetent Elders
Brief Title: Intradermal Influenza Vaccine Study in Elders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); Seattle Institute for Biomedical and Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ID/RD01
Record Dates: First submitted 2007-07-12; First posted 2007-07-19 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Influenza
Keywords: influenza; prevention; intradermal; vaccine; delivery; elderly
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.3 mL Influenza Vaccine ID (Experimental): 60% dose - 0.3 mL delivered intradermally with needle and syringe
  Interventions: Biological: Fluzone Influenza Vaccine (2007-2008)
- 0.15 mL twice Influenza Vaccine ID (Experimental): 60% dose - 0.15 mL delivered twice intradermally with needle and syringe
  Interventions: Biological: Fluzone Influenza Vaccine (2007-2008)
- 0.5 mL Influenza Vaccine by IM (Active Comparator): 100% dose - 0.5mL delivered intramuscularly with needle and syringe
  Interventions: Biological: Fluzone Influenza Vaccine (2007-2008)
- 0.3 mL Influenza Vaccine IM (Experimental): 60% dose - 0.3 mL delivered intramuscularly with needle and syringe
  Interventions: Biological: Fluzone Influenza Vaccine (2007-2008)

INTERVENTIONS:
Biological: Fluzone Influenza Vaccine (2007-2008) — Manufactured by Sanofi Pasteur
  Other Names: Fluzone

SUMMARY:
This randomized trial compared the immunogenicity of 60% dose intradermal (ID) influenza vaccination to standard intramuscular (IM) vaccination of full-dose or 60% dose vaccine. Pre- and postvaccination measurements in the hemagglutination inhibition antibody (HAI) titer were compared. Participants who received reduced-dose vaccine were revaccinated with full-dose IM vaccine.

DETAILED DESCRIPTION:
This study was an open-label randomized trial consisting of community-dwelling adults 65 years and older living in Puget Sound area in Washington State. Subjects were enrolled and randomly assigned to receive licensed, 2007-2008 Northern Hemisphere TIV vaccine (Fluzone, lot U2440AA; Sanofi Pasteur) containing concentrations of hemagglutinin of each of A/Solomon Islands/3/2006 (A/H1N1), A/Wisconsin/67/2005 (A/H3N2), and B/Malaysia/2506/2004 (B): 15 ug/0.5 mL by the IM route, 9 ug/0.3 mL by the ID or IM route, or 4.5 ug/0.15 mL given twice by ID route to the nondominant arm. A block randomization scheme (1:1:1:1), stratified by sex, was used. For IM vaccination, 0.3 mL or 0.5 mL of vaccine was removed from a multidose (5 mL) vial through a 25-gauge, 1-inch detachable needle (Becton Dickinson) and was injected into the deltoid muscle at a 90 degree angle to the skin. For ID vaccination, 0.3 mL or 0.15 mL was drawn by a TB syringe through a 25-gauge, 5/8-inch needle (Terumo Medical). The needle was inserted at a 15 degree angle to the skin overlying the deltoid of the arm. The vaccine was slowly injected until all material was expelled and induration appeared. Subjects randomized to the 0.15-mL group received 2 side-by-side ID injections 3 cm apart. Participants returned at 4 weeks to determine postvaccination antibody titers. At this follow-up visit, those assigned to reduced dose IM or ID influenza vaccinations then received full-dose IM influenza vaccination. These participants returned in another 4 weeks to repeat HAI titers. A nonrandomized subset of subjects (based on availability and willingness to participate) returned at 14 days after initial vaccination for T cell assays in an exploratory substudy to examine cellular immune response.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, medically stable persons 65 years of age or older
* Able to read and understand informed consent
* Available during the trial period and for follow-up
* Able to understand and comply with planned study procedures
* Able to be contacted by telephone for follow-up of adverse events

Exclusion Criteria:

* Known allergy to eggs or other components of vaccine (i.e., thimerosal)
* History of Guillain-Barré Syndrome (GBS)
* Has a confirmed or suspected immunodeficient or immunosuppressive condition (including congenital or acquired immunosuppressive therapy, and human immunodeficiency virus [HIV])
* End-stage renal disease requiring hemodialysis
* Active neoplastic disease or history of any hematologic malignancy (except localized skin or prostate cancer that is stable in the absence of therapy)
* Acute or chronic condition that (in the opinion of the investigator) would render vaccination unsafe or would interfere with the evaluation of responses (including but not limited to the following: known chronic liver disease, significant renal disease, oxygen-dependent chronic lung disease, New York Heart Association Functional Class III or IV, unstable or progressive neurologic disorder, insulin controlled diabetes mellitus)
* Use of experimental vaccines within the month prior to study entry, or expected use of experimental or licensed vaccines or blood/blood products during the duration of the study.
* Receipt of immunoglobulin or other blood product within 3 months prior to enrollment
* Receipt of other licensed vaccines within the preceding 4 weeks
* History of a severe reaction following influenza vaccination
* Current or planned participation in a research study of an investigational drug. Participation in research studies that involve use of licensed drugs, for either approved or investigational indications, will be permitted with the approval of the PI, as will participation in research studies that do not involve vaccines or medications.
* Current use or previous chronic administration, defined as >14 days during the previous six months, of immunosuppressants or other immune-modifying drugs. (For oral or injected corticosteroids, the immune-modifying dose is defined as prednisone or its equivalent >10 mg/day or >800mcg per day of inhaled beclomethasone dipropionate or equivalent ). Topical steroids are allowed.
* Use of cytotoxic therapy in the previous 2 years.
* Plans to receive cytotoxic therapy during the study period.
* Concurrent moderate to severe illness. Need to defer vaccination until recovery. (Vaccination is not contraindicated in subjects with mild illnesses or with low-grade fever).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 257 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Chien Chi, MD, Principal Investigator — VAPSHCS; Kathy Neuzil, MD, Principal Investigator — PATH

REFERENCES:
- [Derived] Chi RC, Rock MT, Neuzil KM. Immunogenicity and safety of intradermal influenza vaccination in healthy older adults. Clin Infect Dis. 2010 May 15;50(10):1331-8. doi: 10.1086/652144. PMID 20377407

RESULTS

PARTICIPANT FLOW:
Groups:
- Full-dose 0.5 mL IM: 0.5 mL influenza vaccine delivered intramuscularly with needle/syringe
- 60% Dose 0.3 mL IM: 0.3 mL influenza vaccine delivered intramuscularly with needle/syringe
- 60% Dose 0.3 mL ID: 0.3 mL influenza vaccine delivered intradermally
- 60% Dose 0.15 mL x 2 ID: 0.15 mL influenza vaccine twice delivered intradermally with needle and syringe
Period: Overall Study
Arm/Group | Full-dose 0.5 mL IM | 60% Dose 0.3 mL IM | 60% Dose 0.3 mL ID | 60% Dose 0.15 mL x 2 ID
Started | 65 | 64 | 64 | 65
Completed | 65 | 64 | 63 | 65
Not Completed | 0 | 0 | 1 | 0
Not completed — Discrepant chart documentation re route | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full-dose 0.5 mL IM | 60% Dose 0.3 mL IM | 60% Dose 0.3 mL ID | 60% Dose 0.15 mL x 2 ID | Total
Number analyzed (Participants) | 65 | 64 | 63 | 65 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 65 | 64 | 63 | 65 | 257
Age Continuous [Mean (Standard Deviation); unit: years] | 75.6 (6.8) | 75.2 (7.7) | 73.6 (6.3) | 74.7 (6.3) | 74.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 11 | 11 | 44
  Male | 54 | 53 | 52 | 54 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 65 | 63 | 62 | 64 | 254
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 3 | 5 | 14
  White | 56 | 60 | 55 | 53 | 224
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 3 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Pre- and Post- Vaccination
Description: Seroprotection before and 4 Weeks after Vaccination by Full- or Reduced-Dose (9 mg) Intramuscular (IM) or Reduced-Dose (9 mg) Intradermal (ID) Injections for A/Solomon Islands/3/2006 (A/H1N1), A/Wisconsin/67/2005 (A/H3N2), B/Malaysia/2506/2004 (B)
Time Frame: 1 month
Measure: Number; unit: % of Participants
Groups:
- Full-dose 0.5 mL IM: 100% dose - 0.5mL delivered intramuscularly with needle and syringe
- 60% Dose 0.3 mL IM: 60% dose - 0.3 mL delivered intramuscularly with needle and syringe
- 60% Dose 0.3 mL ID: 60% dose - 0.3 mL delivered intradermally with needle and syringe
- 60% Dose 0.15 mL x 2 ID: 60% dose - 0.15 mL delivered twice intradermally with needle and syringe
Arm/Group | Full-dose 0.5 mL IM | 60% Dose 0.3 mL IM | 60% Dose 0.3 mL ID | 60% Dose 0.15 mL x 2 ID
Number analyzed (Participants) | 64 | 64 | 63 | 65
% of Participants
  A/H1N1 Seroprotection Prevaccination | 18.5 [34.6 to 66.5] | 12.5 [40.0 to 73.4] | 19.1 | 15.4
  A/H1N1 Seroprotection 4 weeks after vaccination | 65.6 | 57.8 | 68.9 | 67.2
  A/H3N2 Seroprotection Prevaccination | 47.7 | 46.9 | 49.2 | 47.7
  A/H3N2 Seroprotection 4 weeks after vaccination | 76.6 | 75.0 | 75.4 | 75.0
  B Seroprotection Prevaccination | 15.4 | 12.5 | 14.3 | 20.0
  B Seroprotection 4 weeks after vaccination | 26.6 | 17.2 | 16.5 | 25.0

2. Secondary Outcome: Geometric Mean Titer (GMT) Pre- and Post- Vaccination
Description: GMT before and 4 Weeks after Vaccination by Full- or Reduced-Dose (9 mg) IM or Reduced-Dose (9 mg) ID Injections. A/Solomon Islands/3/2006 (A/H1N1), A/Wisconsin/67/2005 (A/H3N2), B/Malaysia/2506/2004 (B)
Time Frame: 1 month
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | Full-dose 0.5 mL IM | 60% Dose 0.3 mL IM | 60% Dose 0.3 mL ID | 60% Dose 0.15 mL x 2 ID
Number analyzed (Participants) | 64 | 64 | 63 | 65
GMT
  A/H1N1 Prevaccination | 12.5 [9.8 to 16.0] | 11.3 [8.9 to 14.3] | 13.6 [10.7 to 17.4] | 11.2 [9.1 to 13.9]
  A/H1N1 4 weeks after vaccination | 54.2 [40.0 to 73.4] | 41.8 [29.5 to 59.2] | 48.0 [34.6 to 66.5] | 48.6 [36.2 to 65.2]
  A/H3N2 Prevaccination | 33.7 [23.9 to 47.6] | 27.1 [20.1 to 36.4] | 29.4 [21.1 to 40.8] | 29.0 [21.2 to 39.7]
  A/H3N2 4 weeks after vaccination | 79.1 [57.6 to 108.6] | 62.4 [46.6 to 83.5] | 57.5 [42.4 to 78.1] | 72.6 [53.2 to 99.1]
  B Prevaccination | 10.7 [8.6 to 13.2] | 10.1 [8.2 to 12.5] | 9.8 [7.8 to 12.3] | 12.8 [9.9 to 16.5]
  B 4 weeks after vaccination | 16.5 [12.7 to 21.4] | 12.4 [10.0 to 15.5] | 10.8 [8.5 to 13.8] | 15.9 [12.1 to 20.9]

3. Secondary Outcome: Assessment of Reactogenicity
Description: Maximum solicited systemic and local signs and symptoms during the week after initial vaccination, by Dose and Randomization Assignment
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | Full-dose 0.5 mL IM | 60% Dose 0.3 mL IM | 60% Dose 0.3 mL ID | 60% Dose 0.15 mL x 2 ID
Number analyzed (Participants) | 64 | 64 | 63 | 65
participants
  Fever, >=38.0C and <39.0C | 0 | 1 | 0 | 3
  Fever, >=39 | 0 | 0 | 0 | 1
  Chills, present but easily tolerated | 1 | 1 | 1 | 6
  Chills, interferes with normal activities | 1 | 1 | 0 | 1
  Fatigue, present but easily tolerated | 4 | 6 | 3 | 8
  Fatigue, interferes with normal activity | 2 | 1 | 0 | 6
  General body ache/pain, present but easily tolerat | 6 | 5 | 3 | 11
  General body ache/pain, interferes with normal a | 1 | 2 | 2 | 4
  Headache, present but easily tolerated | 10 | 5 | 4 | 9
  Headache, interferes with normal activity | 0 | 1 | 0 | 5
  Nausea, present but easily tolerated | 3 | 2 | 2 | 3
  Nausea, interferes with normal activity | 1 | 1 | 0 | 0
  Redness or Discoloration, <=8 cm | 9 | 7 | 45 | 52
  Redness or Discoloration, >8 cm | 0 | 0 | 3 | 4
  Localized swelling, <=8 cm | 13 | 4 | 37 | 44
  Localized swelling, >8 cm | 0 | 0 | 3 | 4
  Pain at injection site, present but easily tolerat | 7 | 11 | 7 | 14
  Pain at injection site, interferes with normal act | 0 | 0 | 0 | 0
  Itching at injection site, present but tolerated | 4 | 5 | 15 | 19
  Itching at injection site, interferes with normal | 0 | 0 | 0 | 2
  Arm motion limitation, some limitiation | 1 | 1 | 0 | 0
  Arm motion limitation, interferes normal activity | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Full-dose 0.5 mL IM | 60% Dose 0.3 mL IM | 60% Dose 0.3 mL ID | 60% Dose 0.15 mL x 2 ID
Serious Adverse Events (participants affected / at risk) | 0/65 | 2/64 | 1/64 | 3/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/64 | 0/64 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full-dose 0.5 mL IM (N=65) | 60% Dose 0.3 mL IM (N=64) | 60% Dose 0.3 mL ID (N=64) | 60% Dose 0.15 mL x 2 ID (N=65)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Resulted in hospitalization.
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Resulted in hospitalization.
anemia and arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Resulted in hospitalization
small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
complicated fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — resulted in hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No